CLINICAL TRIAL: NCT02035657
Title: A Proof-of-Concept Clinical Trial of Intratumoral Injection of GLA-SE, a Toll-like Receptor-4 Agonist, in Patients With Merkel Cell Carcinoma
Brief Title: A Proof-of-Concept Trial of GLA-SE in Patients With Merkel Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immune Design, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDC-G100-2013-001
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Merkel Cell Carcinoma
Keywords: Merkel cell carcinoma; MCC
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — glucopyranosyl lipid-A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GLA-SE (Experimental): Glucopyranosyl Lipid A in Stable Emulsion
  Interventions: Biological: GLA-SE

INTERVENTIONS:
Biological: GLA-SE — Glucopyranosyl Lipid A in Stable Emulsion
  Other Names: Glucopyranosyl Lipid A in Stable Emulsion

SUMMARY:
This is a single arm, open-label, single center study evaluating the safety, feasibility, clinical efficacy and immunogenicity of GLA-SE administration to patients with Merkel cell carcinoma. Ten patients will be treated. The goal is for GLA-SE to assist the patient's own immune system in attacking the cancer cells.

DETAILED DESCRIPTION:
This is a single arm, open-label, single center study evaluating the safety, feasibility, clinical efficacy and immunogenicity of GLA-SE administration to patients with Merkel cell carcinoma. Ten patients with metastatic or locoregional disease will be treated. The goal is for GLA-SE to assist the patient's own immune system in attacking the cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed Merkel cell carcinoma with metastatic or loco-regional disease.
* Patients must have at least one injectable lesion, defined as an easily palpable superficial lesion (cutaneous, subcutaneous or lymph nodal metastasis) that can be accurately localized, stabilized by palpation, and is superficial enough to enable IT injection.
* ECOG performance status score 0, 1 or 2
* ≥ 18 years of age
* Life expectancy of ≥ three months.
* Adequate neutrophil and platelet counts
* Adequate renal and hepatic function
* Willing to undergo pre-treatment lesion biopsy and post-treatment lesion biopsy
* Use of effective contraception
* Signed informed consent document
* Members of all genders, races and ethnic groups are eligible for this trial

Exclusion Criteria:

* Prior chemotherapy or a major surgical procedure within 3 weeks, or radiotherapy within 2 weeks prior to first study treatment
* No concurrent anti-cancer treatment (including topical agents such as imiquimod) or investigational agents
* Active, untreated brain metastases
* Pregnant or nursing
* Use of any systemic immunosuppressive agents
* Immunosuppressed patients
* Uncontrolled depression or other major psychiatric disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility | 1 year
  The number of treatment-related adverse events

SECONDARY OUTCOMES:
Clinical efficacy and Immunogenicity | 1 Year
  The secondary objectives are to assess the clinical efficacy of as well as the immunological effects of GLA-SE in patients with MCC
Clinical efficacy and Immunogenicity | 1 Year
  Objective tumor response rate, time to progression or relapse, survival, and cellular immune activation

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hsu, MD, Study Director — Immune Design, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (1):
- University of Washington Medical Center, Seattle Cancer Care Alliance, Seattle, Washington, United States